CLINICAL TRIAL: NCT00646698
Title: Impact of Body Composition on Very-Low-Density-Lipoprotein-Triglycerides Kinetics
Brief Title: Body Composition and Very-Low-Density-Lipoprotein-Triglycerides (VLDL-TG) Kinetics
Status: Completed | Type: Observational
Sponsor: University of Aarhus (Other)
Collaborators: The Danish Medical Research Council (Other); The Novo Nordic Foundation (Other)
Responsible Party: Soren Nielsen, MD DMsc, Aarhus University Hospital
Other Study IDs: 2004-0217
Record Dates: First submitted 2008-01-07; First posted 2008-03-28 (Estimated); Last update posted 2008-03-28 (Estimated); Status verified 2008-03

CONDITIONS: Obesity; Insulin Resistance
Keywords: VLDL-TG kinetics; Obesity; Body composition; Tracers; Tissue biopsies
MeSH Terms: conditions — Obesity; Insulin Resistance

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- 1: Premenopausal Upper Body Obese (UBO) women with waist-hip ratio > 0.85 and BMI > 28
- 2: Premenopausal Lower Body Obese (LBO) women with waist hip ratio < 0.8 and BMI > 28
- 3: Premenopausal lean women with BMI < 25

SUMMARY:
Context: Upper body obese (UBO) subjects are more likely to develop cardiovascular disease (CVD) than lower body obese (LBO) or lean. This may in part be caused by greater hepatic secretion of very-low-density-lipoprotein-triglycerides (VLDL-TG).

Objective: To assess the impact of body composition and insulin sensitivity on basal VLDL-TG turnover in women.

DETAILED DESCRIPTION:
Body composition is an important predictor of obesity related life-style diseases. Thus, preferential accumulation of adipose tissue in the abdominal region has been demonstrated to be associated with greater risk of developing CVD and insulin resistance than accumulation in lower body depots. The reason for this is not yet fully understood, but there are indications that upper body fat depots contain larger and more lipolytically active adipocytes resulting in an excess hepatic delivery of FFAs in upper body obese individuals. As several lines of experimental evidence as well as cross-sectional studies have demonstrated, elevated levels of FFAs affect the cardiovascular system unfavourably and are most likely a major contributor to insulin resistance. A prominent feature of insulin resistance is hypertriglyceridemia, primarily caused by increased levels of very-low-density-lipoprotein (VLDL)-TG.

Even though lipolysis in subcutaneous adipose tissue accounts for the majority (~75 %) of FFAs delivered to the liver, it is conceivable that excess release from visceral adipocytes in UBO individuals impacts VLDL-TG secretion. The reason for this is two-sided: First, upon entry into the liver, FFAs are reesterified to form VLDL-TG which is subsequently secreted. Studies in cell lines as well as whole body investigations in humans have demonstrated, that perturbations of FFA levels may directly affect VLDL-TG output by the liver. Second, elevated levels of FFAs may induce hepatic insulin resistance resulting in increased VLDL-TG output due to a loss of the inhibitory effect of insulin on VLDL-TG secretion. In theory, this combination of excess substrate availability coupled with an unfavorable hormonal milieu (hepatic insulin resistance) could result in increased VLDL-TG production in UBO subjects. A recent study by Mittendorfer et. al. support this notion, since weight loss in UBO women resulted in decreased VLDL-TG production, presumably caused primarily by a decrease in the supply of visceral fatty acids.

Although findings from previous studies have been contradictory as to whether body fat distribution directly affects VLDL-TG clearance, in vitro findings suggest regional differences in lipoprotein lipase (LPL) activity between UBO and LBO women, and VLDL-TG clearance could also be modulated by differences in VLDL associated fatty acid oxidation. To our knowledge, the latter point has not previously been addressed.

The purpose of this study was therefore to investigate differences in VLDL-TG kinetics in women with different body composition phenotypes. Our preliminary hypothesis was that UBO women produce and secrete greater amounts of VLDL-TG than their lower body obese (LBO) or lean counterparts. We also hypothesized, that peripheral clearance would be similar in all groups. Lastly, we wanted to investigate whether the more benevolent lipid profile seen in lean women could in part be a result of a more efficient channeling of VLDL derived fatty acids towards oxidation.

ELIGIBILITY:
Inclusion Criteria:

* Woman
* Premenopausal
* Healthy
* Not taking medication

Exclusion Criteria:

* Diabetes

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Community sample
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2006-04; Primary Completion 2007-02 (Actual); Study Completion 2007-06 (Actual)

PRIMARY OUTCOMES:
VLDL-TG kinetics were assessed using a bolus injection of ex-vivo labeled [1-14C]VLDL-TG | Hours

SECONDARY OUTCOMES:
fractional VLDL-TG derived fatty acid oxidation was measured by 14CO2 trapping from expired air | Hours
VLDL-TG fat deposition by adipose tissue biopsies | Hours
Insulin sensitivity by the hyperinsulinemic-euglycemic clamp technique | 2 hours

CONTACTS AND LOCATIONS:
Overall Officials: Lars C Gormsen, MD PhD, Principal Investigator — Aarhus University Hospital, Department M
Locations (1):
- Medical Research Laboratories, Aarhus, Denmark